CLINICAL TRIAL: NCT01782963
Title: A Phase II Study of Modified Lenalidomide, Bortezomib and Dexamethasone for Transplant-Ineligible Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Lenalidomide/Bortezomib/Dexamethasone for Multiple Myeloma (MM)
Acronym: RVD Lite
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Noopur Raje, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-498
Record Dates: First submitted 2013-01-15; First posted 2013-02-04 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Multiple Myeloma
Keywords: Newly diagnosed
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Induction (Cycles 1-9): Lenalidomide orally, days 1-21. Bortezomib injection, days 1, 8, 15, 22. Dexamethasone orally, days 1, 2, 8, 9, 15, 16, 22, 23 (for subjects 75 years of age or younger), or Dexamethasone orally days 1, 8, 15, 22 (for subjects greater than 75 years of age)
  Consolidation (cycles 10-15): Lenalidomide po daily (1-21). Bortezomib sc on days 1, 15
  Interventions: Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide
  Other Names: Revlimid
Drug: Bortezomib
  Other Names: Velcade
Drug: Dexamethasone

SUMMARY:
This research study is a Phase II clinical trial. Phase II clinical trials test the effectiveness of an investigational combination of drugs. The purpose is to learn whether the combination of drugs works in treating a specific cancer. "Investigational" means that the combination of drugs is still being studied. It also means that research doctors are trying to find out more about it. Examples of what they want to learn about are the safest dose to use, the side effects it may cause, and if the combination of drugs works for treating different types of cancer.

DETAILED DESCRIPTION:
If you are willing to participate in this study you will be asked to undergo some screening procedures and tests to confirm that you are eligible. Many of these tests and procedures are likely to be part of regular cancer care. They may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated. These tests and procedures include: a medical history, physical exam, performance status, vital signs, neurological exam, bone imaging studies, chest x-ray, bone marrow aspirate, ECG, blood tests and urine tests. If these tests show that you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in the research study.

For cycles 1-9 (each cycle lasts 35 days) you will receive the following: Lenalidomide-once a day on Days 1-21. You will take Lenalidomide by mouth at the same time each day. Bortezomib- once a day on Days 1, 8, 15 and 22. If you are one of the first ten patients enrolled you will get Bortezomib as an intravenous injection for the first cycle. You will get Bortezomib as an injection under the skin for all other cycles. If you are not one of the first 10 patients enrolled you will get Bortezomib as an injection under the skin for all cycles. Dexamethasone-if you are 75 years old or younger you will get Dexamethasone on Days 1, 2, 8, 9, 15, 16, 22 and 23. If you are more than 75 years old you will get Dexamethasone on Days 1, 8, 15 and 22. You will take Dexamethasone by mouth at the same time each day.

For cycles 10-15 (each cycle lasts 28 days) you will receive the following: Lenalidomide-once a day on Days 1-21. You will take Lenalidomide by mouth at the same time each day. Bortezomib-Once a day on Days 1 and 15. You will get Bortezomib as an injection under the skin. You will be given a drug diary to record taking your doses of the drugs. The study staff will tell you how to complete the diary.

During the study you will have to come to the clinic for visits. The tests and procedures that will be done at each visit are listed below:

Day 1 of all cycles: questions about health, medications etc., physical exam, performance status, vital signs, neurological exam, questionnaires, bone imaging studies, bone marrow aspirate, blood tests, pregnancy test, education and counseling, collection of bone marrow, plasma and serum (cycle 1 only), urine test.

Day 8 of cycles 1-9: questions about health, medications etc., vital signs, blood tests.

Day 15 of all cycles: questions about health, medications, etc., vital signs, blood tests, pregnancy test.

Day 22 of cycles 1-9: questions about health, medications, etc., vital signs, blood tests.

After the final dose of the study drug you will have an End of Treatment visit. The following tests and procedures will be done at this visit: questions about health, medications etc., physical exam, performance status, vital signs, neurological exam, questionnaires, bone imaging studies, bone marrow aspirate, blood tests, pregnancy test, education and counseling, collection of bone marrow, plasma and serum, urine test.

After your End of Treatment visit, we would like to follow your status every 2 months until your disease gets worse. The following tests and procedures will be done at these follow-up visits: questions about health, medications, symptoms etc., blood tests and urine test.

If you are one of the first twenty patients enrolled in the study you will also be asked to provide additional blood samples to study what the body does to the study drug. We will take one sample at five time points during cycle 1 and 2. Collection of these samples may require you to come back into the clinic on additional days when you are not receiving study drugs.

You will be in this research study for about 15 months. You can be in this study for a maximum of 15 cycles. If your disease gets worse before the 15th cycle you will be taken off the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented symptomatic myeloma, with organ damage related to myeloma
* Myeloma that is measurable either by serum or urine evaluation of the monoclonal component or by assay of serum free light chains
* Must commit to complete abstinence from heterosexual contact or begin two acceptable method of birth control, one highly effective method and one additional effective (barrier) method

Exclusion Criteria:

* Eligible for autologous stem cell transplantation
* HIV positive on combination antiretroviral therapy
* Pregnant or breastfeeding
* Treated with any prior systemic therapy
* Primary amyloidosis or myeloma complicated by amyloidosis
* Receiving other investigational agents within 14 days of the start of this trial or during this trial
* Known brain metastases
* Poor tolerability or known allergy to any of the study drugs or similar compounds
* Intercurrent illness
* Previous history of another malignant condition except for basal cell carcinoma or stage I cervical cancer
* Inability to comply with an anti-thrombotic treatment regimen
* Peripheral neuropathy greater than or equal to grade 2

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - John Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital/North Shore Cancer Center, Danvers, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: Induction (Cycles 1-9): Lenalidomide orally, days 1-21. Bortezomib injection, days 1, 8, 15, 22. Dexamethasone orally, days 1, 2, 8, 9, 15, 16, 22, 23 (for subjects 75 years of age or younger), or Dexamethasone orally days 1, 8, 15, 22 (for subjects greater than 75 years of age)
  Consolidation (cycles 10-15): Lenalidomide po daily (1-21). Bortezomib sc on days 1, 15
  Lenalidomide
  Bortezomib
  Dexamethasone
Period: Overall Study
Arm/Group | Treatment Arm
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 73 [65 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42
  Black or African-American | 2
  Asian | 3
  Other | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50
ISS Stage at Diagnosis [Count of Participants; unit: Participants] — International Staging System for Multiple Myeloma, divides multiple myeloma into three categories with III representing more advanced disease and I less advanced disease
  Stage I :
  * Serum beta-2 microglobulin is less than 3.5 mg/L
  * AND Albumin level is 3.5 g/dL or greater
  * AND Cytogenetics are considered "not high risk"
  * AND Lactate dehydrogenase (LDH) levels are normal
  Stage II: Not stage I or stage II
  Stage III:
  * Serum beta-2 microglobulin is 5.5 (mg/L) or greater
  * AND Cytogenetics are considered "high-risk"
  * AND/OR LDH levels are high
  Participants
    I | 19
    II | 17
    III | 14
Durie-Salmon Stage [Count of Participants; unit: Participants] — Stage III represents more advanced disease and stage I less advanced.
  Stage I:
  * Hemoglobin value 10 g/dL
  * Serum calcium value normal or =12 mg/dL
  * Bone x-ray, normal bone structure (scale 0) or solitary bone plasmacytoma only
  * Low M-component production rate (IgG value <5 g/dL; IgA value <3 g/dL; Bence Jones protein <4 g/24 hr)
  Stage II:
  Neither stage I nor stage III
  Stage III:
  On or more of the following:
  * Hemoglobin value 12 mg/dL
  * Advanced lytic bone lesions (scale 3)
  * High M-component production rate - IgG value >7 g/dL; IgA value>5 g/dL; Bence Jones protein >12 g/24 h
  Participants
    I | 16
    II | 16
    III | 18
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Performance Status Score
  * 0: Asymptomatic (Fully active, no restrictions in self care)
  * 1: Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature)
  * 2: Symptomatic, <50% time in bed during the day (Ambulatory and capable of all self care but unable to carry out any work activities)
  * 3: Symptomatic, >50% time in bed during waking hours (Capable of only limited self-care)
  * 4: Bedbound (Completely disabled. Cannot carry on any self-care)
  * 5: Death
  Participants
    0 | 25
    1 | 18
    2 | 7
    3 | 0
    4 | 0
    5 | 0
High-Risk Cytogenetics [Count of Participants; unit: Participants] — Cytogenetics risk is determined by doing a genetic analysis of the participants bone marrow. The participants chromosomes are assessed for things like translocations (rearrangement of non-homologous chromosomes) or deletions (part of the genetic sequence is lost). Participants were considered high-risk if they had certain specific genetic changes. Translocations are noted as t(chromosome 1; chromosome 2) where the two chromosomes represent which non homologous chromosomes swapped genetic material. The high-risk cytogenetics included a deletion on chromosome 17, t(4;14), t(14;16), and t(14;20).
  Participants
    Yes | 6
    No | 42
    Unknown | 2
Serum Heavy/Light Chain [Count of Participants; unit: Participants] — The serum heavy/light chain immunoassay quantifies the light chain types of each immunoglobulin (Ig) class based on a sample of the participants blood. Typical antibodies consist of two Ig heavy chains connected to two Ig light chains. When the plasma cells become cancerous, it can result in an increase in monoclonal immunoglobulin in the blood serum. This is used as a measure of the tumor load. The information below gives which specific monoclonal immunoglobulin was detected.
  Participants
    IgG | 34
    IgA | 9
    Light-chain only | 5
    Unknown | 2
Body Mass Index (BMI) [Median (Full Range); unit: Kg/m^2] | 28 [18 to 45]

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Participants are considered to have achieved an objective response if they meet the International Myeloma Working Group uniform response criteria for any of the following:
  * Stringent CR: Same as CR plus normal free light chain ratio and absence of clonal cells plasma cells in bone marrow (BM)
  * CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in BM
  * VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100 mg per 24 hours
  * PR: ≥50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ≥90% or to <200 mg per 24 hours. If the serum and urinary M-protein are not measurable, additional criteria are used to assess PR that will not fit in the space provided here. If present at baseline, a ≥50% reduction in the size of plasmacytomas is also required
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 50
Participants
  Stringent Complete Response | 6
  Complete Response (CR) | 16
  Very Good Partial Response (VGPR) | 11
  Partial Response (PR) | 10

2. Secondary Outcome: Number of Participants With Grade 3 or Higher Treatment Related Adverse Events
Description: A summary of the number of participants with grade 3 or higher treatment related adverse events for adverse events that had an overall incidence of greater than 15% (any grade) as assessed by Common Terminology Criteria for Adverse Events (CTCAE 4).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 50
Participants
  Fatigue | 8
  Peripheral Neuropathy | 1
  Hypophosphatemia | 17
  Neutropenia | 7
  Diarrhea | 0
  Peripheral Edema | 1
  Insomnia | 1
  Rash | 5
  Anemia | 1
  Thrombocytopenia | 1
  Constipation | 0
  Dysgeusia | 0
  Hyperglycemia | 2
  Nausea | 0
  Depression | 0
  Psychiatric Disorder, other | 2
  Generalized Muscle Weakness | 2

3. Secondary Outcome: Median Progression Free Survival
Description: The median amount of time as measured from the start of treatment until either death or progression.
  Progressive disease requires 1 or more of the following:
  * >=25% increase from lowest response level in serum M-protein (>=0.5 g/dL absolute increase) and/or urine M-component (>=200 mg/24hr absolute increase)
  * >=25% increase in the difference between involved and uninvolved FLC levels (absolute increase >10 mg/dL). Only for use in patients without measurable serum and M-protein levels.
  * >=25% increase in bone marrow plasma cell percentage (absolute percentage >=10%)
  * New or increase in existing bone lesions or soft tissue plasmacytomas
  * Hypercalcemia (serum calcium >11.5 mg/dL) due solely to the plasma cell proliferative disorder.
Time Frame: From the start of treatment until death or progression or until 3 years after the last participant is enrolled
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 50
Months | 35.1 [30.9 to NA] — Upper bound is infinity due to skew of survival data

4. Secondary Outcome: Median Overall Survival
Description: The median overall survival as measured from the start of treatment until the time of death due to any cause.
Time Frame: From the start of treatment until death or until 5 years after the time of disease progression
Population: Median overall survival was not met before the end of follow-up/ data cutoff point because more than half of the participants were still alive.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Treatment Arm
Number analyzed (Participants) | 50
years | NA [NA to NA] — Median overall survival was not met before the data cutoff point because more than half of the participants were still alive

5. Secondary Outcome: Median Time to Response
Description: Median amount of time from the start of treatment until first documented response as defined by the International Myeloma Working Group uniform response criteria
  Stringent CR: Same as CR plus normal free light chain ratio and absence of clonal cells plasma cells in bone marrow (BM) CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in BM VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100 mg per 24 hours PR: ≥50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ≥90% or to <200 mg per 24 hours. If the serum and urinary M-protein are not measurable, additional criteria are used to assess PR that will not fit in the space provided here. If present at baseline, a ≥50% reduction in the size of plasmacytomas is also required
Time Frame: From the start of treatment until the time of first documented response, median duration of 1.1 months
Population: Participants that achieved a response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 43
Months | 1.1 [1.1 to 1.3]

6. Secondary Outcome: Response Rate With Respect to Cytogenetic Characteristics
Description: Response rate was assessed using the International Myeloma Working Group uniform response criteria. Stringent complete response, Complete Response, Very Good Partial Response, and Partial Response are defined in outcome measure 1.
  * MR included participants in whom some, but not all, criteria for PR were fulfilled, providing the remaining criteria satisfied the requirements for MR. Required all of the following:
    * ≥25% to ≤ 49% reduction in the level of serum monoclonal protein for at least two determinations six weeks apart.
    * If present, a 50 to 89% reduction in 24-hour light chain excretion, which still exceeds 200 mg/24 h, for at least two determinations six weeks apart.
    * 25-49% reduction in the size of plasmacytomas (by clinical or radiographic examination) for at least six weeks.
    * No increase in size or number of lytic bone lesions (development of compression fracture does not exclude response).
  * Stable Disease: Not meeting the criteria for minimal response or
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- High Risk Cytogenetics; Low Risk Cytogenetics: Induction (Cycles 1-9): Lenalidomide orally, days 1-21. Bortezomib injection, days 1, 8, 15, 22. Dexamethasone orally, days 1, 2, 8, 9, 15, 16, 22, 23 (for subjects 75 years of age or younger), or Dexamethasone orally days 1, 8, 15, 22 (for subjects greater than 75 years of age)
  Consolidation (cycles 10-15): Lenalidomide po daily (1-21). Bortezomib sc on days 1, 15
  Lenalidomide
  Bortezomib
  Dexamethasone
Arm/Group | High Risk Cytogenetics | Low Risk Cytogenetics
Number analyzed (Participants) | 6 | 44
Participants
  Stringent Complete Response | 0 | 6
  Complete Response | 2 | 14
  Very Good Partial Response | 2 | 9
  Partial Response | 1 | 9
  Minimal Response | 1 | 0
  Stable Disease | 0 | 3
  Not evaluable | 0 | 3

7. Secondary Outcome: Mean Plasma Bortezomib Concentration Following Intravenous and and Subcutaneous Injection
Description: The pharmacokinetic profile of intravenous and subcutaneous bortezomib administration in combination with lenalidomide and dexamethasone.
Time Frame: Day 1 (5 min, 30min, 5 hours post dose), Days 8, 15, Day 22 (pre dose and 5 min, 30 min, 5 hrs post dose), cycle 2 day 1 pre dose
Population: A total of only 10 participants per arm were evaluated for drug plasma concentrations following Bortezomib administration.The number of participants vary by time-point due to missing measurements for the concentrations.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Intravenous: Induction (Cycles 1-9): Lenalidomide orally, days 1-21. Bortezomib injection, days 1, 8, 15, 22. Dexamethasone orally, days 1, 2, 8, 9, 15, 16, 22, 23 (for subjects 75 years of age or younger), or Dexamethasone orally days 1, 8, 15, 22 (for subjects greater than 75 years of age)
  Consolidation (cycles 10-15): Lenalidomide po daily (1-21). Bortezomib sc on days 1, 15
  Lenalidomide
  Bortezomib
  Dexamethasone
- Subcutaneous: Induction (Cycles 1-9): Lenalidomide orally, days 1-21. Bortezomib injection, days 1, 8, 15, 22. Dexamethasone orally, days 1, 2, 8, 9, 15, 16, 22, 23 (for subjects 75 years of age or younger), or Dexamethasone orally days 1, 8, 15, 22 (for subjects greater than 75 years of age)
  Consolidation (cycles 10-15): Lenalidomide po daily (1-21). Bortezomib sc on days 1, 15
  Lenalidomide
Arm/Group | Intravenous | Subcutaneous
Number analyzed (Participants) | 10 | 10
ng/mL
  Day 1, 5 minutes (min) post dose | 98.84 (39.27) | 13 (15.79)
  Day 1, 30 min post dose | 8.73 (5.59) | 20.5 (10.91)
  Day 1, 5 hours post dose: number analyzed (Participants) | 10 | 9
  Day 1, 5 hours post dose | 1.82 (1.31) | 1.96 (0.56)
  Day 8 pre-dose | 0.44 (0.15) | 0.33 (0.09)
  Day 15 pre-dose: number analyzed (Participants) | 8 | 10
  Day 15 pre-dose | 0.66 (0.22) | 0.49 (0.12)
  Day 22 pre-dose: number analyzed (Participants) | 7 | 9
  Day 22 pre-dose | 0.83 (0.34) | 0.66 (0.18)
  Day 22, 5 min post-dose: number analyzed (Participants) | 7 | 9
  Day 22, 5 min post-dose | 114.3 (76.6) | 10.29 (13.24)
  Day 22, 30 min post-dose: number analyzed (Participants) | 7 | 9
  Day 22, 30 min post-dose | 14.9 (4.3) | 21.69 (10.1)
  Day 22, 5 hours post-dose: number analyzed (Participants) | 7 | 9
  Day 22, 5 hours post-dose | 2.85 (1.05) | 4.16 (2.07)
  Cycle 2 Day 1, pre-dose: number analyzed (Participants) | 9 | 9
  Cycle 2 Day 1, pre-dose | 0.53 (0.15) | 0.49 (0.14)

8. Secondary Outcome: Pharmacogenomic Markers of Neuropathy
Description: To evaluate pharmacogenomic markers among patients with treatment related polyneuropathy.
Time Frame: 2 years
Population: No pharmacogenomic markers were evaluated for relation to neuropathy
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the end of treatment (approximately 16 months)
Description: Serious adverse events were defined as any grade 3 or greater adverse event that was deemed to be at least potentially related to one of the study drugs.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 34/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=50)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Corneal ulcer (Eye disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Eye disorders - Other, Sclera redness (Eye disorders) | 1 (1)
Fatigue (General disorders) | 8 (9)
Gastrointestinal disorders - Other, Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, GI Bleed (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Heart failure (Cardiac disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 15 (20)
Hypotension (Vascular disorders) | 1 (2)
Nervous system disorders - Other, Altered mental status and loss of consciousness (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=50)
Abdominal distension (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 5 (7)
Agitation (Psychiatric disorders) | 5 (7)
Alanine aminotransferase increased (Investigations) | 5 (6)
Alkaline phosphatase increased (Investigations) | 5 (14)
Anemia (Blood and lymphatic system disorders) | 30 (62)
Anorexia (Metabolism and nutrition disorders) | 12 (17)
Anxiety (Psychiatric disorders) | 8 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 7 (9)
Atrial fibrillation (Cardiac disorders) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (30)
Blood bilirubin increased (Investigations) | 3 (14)
Blurred vision (Eye disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (8)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Confusion (Psychiatric disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 22 (30)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Creatinine increased (Investigations) | 4 (16)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Depression (Psychiatric disorders) | 11 (12)
Diarrhea (Gastrointestinal disorders) | 25 (37)
Dizziness (Nervous system disorders) | 10 (11)
Dry mouth (Gastrointestinal disorders) | 6 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6)
Dysgeusia (Nervous system disorders) | 13 (17)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (22)
Edema face (General disorders) | 4 (6)
Edema limbs (General disorders) | 23 (37)
Fatigue (General disorders) | 41 (92)
Fever (General disorders) | 5 (5)
Flu like symptoms (General disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 10 (11)
Headache (Nervous system disorders) | 6 (6)
Hearing impaired (Ear and labyrinth disorders) | 4 (4)
Hot flashes (Vascular disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 20 (33)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (5)
Hypertension (Vascular disorders) | 20 (72)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (20)
Hypokalemia (Metabolism and nutrition disorders) | 10 (13)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (13)
Hyponatremia (Metabolism and nutrition disorders) | 13 (26)
Hypophosphatemia (Metabolism and nutrition disorders) | 27 (68)
Hypotension (Vascular disorders) | 8 (11)
INR increased (Investigations) | 3 (4)
Insomnia (Psychiatric disorders) | 19 (23)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 10 (11)
Neutrophil count decreased (Investigations) | 7 (23)
Non-cardiac chest pain (General disorders) | 3 (4)
Oral pain (Gastrointestinal disorders) | 3 (3)
Pain (General disorders) | 12 (23)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (26)
Pelvic pain (Reproductive system and breast disorders) | 4 (4)
Peripheral motor neuropathy (Nervous system disorders) | 7 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 32 (59)
Platelet count decreased (Investigations) | 16 (48)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16 (35)
Rhinitis infective (Infections and infestations) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 8 (21)
Spinal fracture (Injury, poisoning and procedural complications) | 4 (4)
Thromboembolic event (Vascular disorders) | 5 (6)
Upper respiratory infection (Infections and infestations) | 15 (22)
Urinary tract infection (Infections and infestations) | 7 (8)
Vomiting (Gastrointestinal disorders) | 6 (8)
Weight loss (Investigations) | 8 (8)
White blood cell decreased (Investigations) | 13 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No